CLINICAL TRIAL: NCT06263543
Title: SERIES: SEquencing Sacituzumab Govitecan AfteR T-DXd In ER+/HER2 LOW/ULTRA LOW MetaStatic Breast Cancer
Brief Title: Sequencing Antibody Drug Conjugates in ER+/HER2 LOW/ULTRA LOW MBC
Acronym: SERIES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reshma L. Mahtani, D.O. (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Reshma L. Mahtani, D.O., Chief of Breast Medical Oncology, Baptist Health South Florida
Organization: Baptist Health South Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-MAH-001
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Hormone-receptor-positive Breast Cancer; Human Epidermal Growth Factor 2 Low Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan (SG) Infusion (Experimental): SG will be administered on Days 1 and 8 of continuous 21-day cycles at 10 mg/kg via intravenous (IV) infusion until disease progression or unacceptable toxicity.
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — IV infusion of 10 mg/kg on Days 1 and 8 of each continuous and consecutive 21-day cycles. The first infusion will last approximately 3 hours and subsequent infusions will last 1-2 hours if prior infusions were well tolerated.
  Other Names: Trodelvy

SUMMARY:
The purpose of this research study is to see if the medication sacituzumab govitecan (SG) is effective at the currently approved dose and schedule in people who have previously received trastuzumab deruxtecan (T-DXd) for the treatment of metastatic, hormone receptor positive (HR+)/human epidermal growth factor 2 low (HER2 low) breast cancer. Although SG is approved to treat metastatic HR+/HER2 negative breast cancer, the aim of this study is to determine if SG is still effective specifically in people who have already received T-DXd.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Individuals ≥ 18 years of age.
* 4. Histologically confirmed metastatic or advanced and unresectable breast cancer that is HER2 LOW/ULTRA LOW by local testing on either the primary or any metastatic site. HER2 LOW is defined as: (IHC 2+/ISH- or IHC 1+ (ISH- or untested)) and HER2 ULTRA LOW is defined as: IHC0+ (faint membrane staining up to 10%)
* Histologically confirmed metastatic or advanced and unresectable breast cancer that is hormone receptor positive (estrogen receptor and/or progesterone receptor positive) defined as >1% on any metastatic site or the primary tumor.
* Endocrine-refractory (as per investigator judgement) and may have received any number of prior endocrine therapies (alone or in combination with cyclin-dependent kinase (CDK)4/6 inhibitor, everolimus, alpelisib, acapivasertib or inavolisib).
* Received a CDK4/6 inhibitor either alone or in combination with endocrine therapy (in the adjuvant or metastatic setting) with any duration of therapy permitted.
* Received at least 1 but no more than 4 prior systemic chemotherapy regimens in the metastatic setting. Prior ADCs count as a line of systemic chemotherapy. Prior PARP inhibitor use counts as a line of systemic therapy.
* Prior treatment with T-DXd (discontinued for progression and/or intolerance), which does not have to be the treatment immediately prior to enrollment on trial.
* Documented clinical and/or radiographic disease progression after most recent therapy, unless immediate prior therapy was T-DXd which was discontinued for toxicity.
* Measurable disease, as per RECIST V1.1 - a. If a patient has bone-only disease, they are eligible as long as there is a lytic lesion that is considered measurable. Blastic-only bone lesions are not allowed.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2.
* Adequate organ and bone marrow function within 28 days before enrollment. For all parameters listed below, the most recent results available must be used:

  1. Hemoglobin ≥ 9 g/dL. Note: Red blood cell transfusion is not allowed within 1 week prior to screening assessment.
  2. Absolute neutrophil count (ANC) ≥ 1500/mm^3. Note: Granulocyte-colony stimulating factor (G-CSF) administration is not allowed within 1 week prior to screening assessment.
  3. Platelet count ≥ 100,000/mm^3. Note: Platelet transfusion is not allowed within 1 week prior to registration.
  4. Total bilirubin (TBL) ≤ 1.5 × upper limit of normal (ULN) if no liver metastases or < 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastasis at baseline.
  5. Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 ×ULN or < 5 × ULN in patients with liver metastasis.
  6. Serum albumin ≥ 2.5 g/dL.
  7. Creatinine clearance (CrCl) ≥ 30 mL/min (calculated using the Cockcroft and Gault equation). Cockcroft-Gault equation: CrCl (mL/min) = [140 - age (years)] × weight (kg) 72 × serum creatinine (mg/dL) {× 0.85 for females}
  8. International normalized ratio (INR) or prothrombin time (PT) and either partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
* Adequate treatment washout period before randomization, defined as:

  1. Major surgery: ≥ 3 weeks
  2. Radiation therapy including palliative and/or stereotactic radiation therapy ≥ 2 weeks
  3. Hormonal therapy: ≥ 2 weeks
  4. Targeted therapy (CDK4/6i, PARP inhibitor, AKTinhibitor, mTOR inhibitor, PIK3CA inhibitor): ≥ 2 weeks
  5. Immunotherapy (non-antibody-based therapy): ≥ 2 weeks
  6. T-DXd: ≥ 3 weeks
* Evidence of post-menopausal status or for individuals of childbearing potential must have a negative serum beta-human chorionic gonadotropin (ß-hCG) at screening or baseline. Individuals of childbearing potential are defined as those who are not surgically sterile (i.e., underwent bilateral tubal occlusion, bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal.
* Individuals of childbearing potential who are sexually active with a non-sterilized male partner must agree to use at least one highly effective method of contraception from the time of registration through final study treatment. Not all methods of contraception are highly effective.
* Non-sterilized male patients who are sexually active with a partner of childbearing potential must agree to use a condom with spermicide from registration and throughout duration of the study treatment.

The following are acceptable measures to prevent pregnancy:

* Abstinence (not having sexual relations with a person who can get you pregnant)
* Non-hormonal Intrauterine Device (IUD)
* Vasectomy
* Sterilization
* Bilateral tubal occlusion

Exclusion Criteria:

* Locally advanced MBC (stage IIIc) in individuals who are candidates for curative intent therapy at the time of study enrollment.
* Patients with brain metastases (BM) except for asymptomatic treated BM not requiring ongoing corticosteroid treatment with stable lesions on baseline/screening brain MRI. Patients who require treatment of brain metastases are eligible after 14 days post receipt of surgery or radiation, if felt to be clinically stable and not requiring ongoing corticosteroid treatment.
* Active serious infection requiring ongoing antibiotics.
* History of an anaphylactic reaction to irinotecan.
* Pregnant or breastfeeding.
* Ongoing treatment with another investigational drug or other interventional trial.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Any other condition that may put a participant at higher risk, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 24 months
  ORR will be assessed using Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1). ORR is defined as the percentage of participants who received at least one dose of SG and have achieved a complete response (CR) or partial response (PR) as assessed by the local investigator.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | 24 months
  CBR will be assessed using RECIST 1.1 and is defined as the percentage of participants who received at least one dose of SG and have achieved CR, PR, or stable disease (SD) as assessed by the local investigator.
Progression-free survival (PFS) | 30 months
  PFS is defined as the duration of time from the date of first treatment until the date of the first radiological progressive disease (PD) per RECIST 1.1 or death from any cause, whichever comes first.
Overall survival (OS) | 30 months
  OS is defined as the duration of time of first treatment until the date of death from any cause.
Duration of response (DOR) | 30 months
  DOR is defined as the duration of time from the date of first response (CR or PR) until the date of the first radiological PD per RECIST 1.1 or death from any cause, whichever comes first.
Global Quality of Life | 24 months
  Global Quality of Life is measured by European Organisation for Research and Treatment of Cancer Core Questionnaire (EORTC QLQ-C30), a 30-item instrument designed to measure quality of life in individuals with cancer. The items are related to how difficult activities of daily living are, how often treatment or cancer-related symptoms occur and how much they interfere in daily activities and relationships. Each item is scored on a scale of 1 (not at all) to 4 (very much). Higher scores indicate worse quality of life.
Treatment-related Adverse Events (AEs) and Serious Adverse Events (SAEs) | 30 months
  Percent of participants who experienced a treatment-related AE or SAE while on study.
Laboratory and Vital Sign Abnormalities | 30 months
  Percent of participants who experienced a laboratory or vital sign abnormality that was considered clinically significant by the investigator while on study.
Growth Factor Support | 30 months
  Percent of participants who required the use of growth factor support (administered at the discretion of the investigator) while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma L Mahtani, D.O., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (3):
- United States (3):
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rugo HS, Bardia A, Tolaney SM, Arteaga C, Cortes J, Sohn J, Marme F, Hong Q, Delaney RJ, Hafeez A, Andre F, Schmid P. TROPiCS-02: A Phase III study investigating sacituzumab govitecan in the treatment of HR+/HER2- metastatic breast cancer. Future Oncol. 2020 Apr;16(12):705-715. doi: 10.2217/fon-2020-0163. Epub 2020 Mar 30. PMID 32223649
- [Background] Schmid P, Cortés J, Marmé F, Rugo HS, Tolaney SM, Oliveira M, Loirat D, Jhaveri K, Yoon OK, Motwani M, Wang H, Delaney RJ, Bardia A. Sacituzumab govitecan (SG) efficacy in hormone receptor-positive/human epidermal growth factor receptor 2-negative (HR+/HER2-) metastatic breast cancer (MBC) by HER2 immunohistochemistry (IHC) status in the phase III TROPiCS-02 study. Annals of Oncology. 2022; 33(Suppl7): S635-636.
- See also: Miami Cancer Institute — https://cancer.baptisthealth.net/